CLINICAL TRIAL: NCT06787092
Title: The Outcome of Pre-transplant Bladder Cycling in Patients With Defunctionalized Bladder
Acronym: PBC and DF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Shaker, assistant lecturer, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bladder cycling
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cycling, Defunctionalized Bladder
Keywords: bladder cycling, defunctionalized bladder

STUDY DESIGN:
Intervention Model Description: the study main objective is to describe various parameters related to bladder functionality in renal transplanted cases with defunctionalized bladder when treated with pre-transplant bladder cycling and due to limited data available, estimation of sample size will be based on effect size. A sample size of at least 20 cases achieves a power of 80% to detect a large effect size of 0.7 comparing pre- and post- cystometric capacity using paired t-test with level of significance of 0.05.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Egyptian patients attending Ain Shams University hospitals (Experimental): ESRD patients maintained on hemodialysis for more than 12 months having oliguria or anuria with reduced bladder capacity (less than 100 ml) assessed by cystogram.
  Interventions: Procedure: bladder cycling

INTERVENTIONS:
Procedure: bladder cycling — started by the instillation of the sterile water in the bladder in amount equal to the estimated bladder capacity. Then the amount will be gradually increased till the patient can withstand filling the bladder with 250 cc of sterile saline for 2 hours.

SUMMARY:
The aim of this study is to evaluate the efficacy of pre-transplant programmed bladder cycling for patient with defunctionalized urinary bladder

DETAILED DESCRIPTION:
Kidney transplantation still remains the best treatment for end-stage renal disease (ESRD). Indeed, increasing numbers of patients are referred for transplantation, but there has been no concomitant increase in the supply of kidneys from the traditional donor pool. Many potential recipients awaiting transplantation, therefore must undergo dialysis for a long time. Regarding the detrimental effect of long-term dialysis associated with oliguria or anuria on the lower urinary tract, and especially in bladder, the interruption of physiological cycle of storage and voiding brings to a situation called Defunctionalized Bladder (DB) in which the bladder capacity became smaller in size. (Errando et al 2018).

In this study we will evaluate the outcome of renal transplantation into a defunctionalized bladder by comparing direct transplantation into this defunctionalized bladder and pre-transplant programmed bladder cycling.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 16 years and older.
2. ESRD patients maintained on hemodialysis for more than 12 months.
3. Have oliguria or anuria
4. reduced bladder capacity (less than 100 ml) assessed by cystogram.

Exclusion Criteria:

* 1- Previous bladder or pelvic surgery or procedure having affected the bladder function.

  2- Neurogenic bladder dysfunction. 3-Patients with history of lower urinary tract symptoms before developing renal failure.

  4-Those with lower urinary tract disease resulting in renal failure.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
measuring bladder size | 3 months
  measuring bladder size by ACUG

SECONDARY OUTCOMES:
increasing bladder size to facilitate uretrovesical reimplantation during renal transplantationn | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all my IPD can be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: will be available at any time forever
Access Criteria: medical student only

REFERENCES:
- [Result] Silverii H, Cain MP. A novel approach to bladder cycling for defunctionalized bladders prior to pediatric kidney transplantation: A case series. J Pediatr Urol. 2024 Aug;20(4):762-764. doi: 10.1016/j.jpurol.2024.03.022. Epub 2024 Mar 24. PMID 38570243
- [Result] Osman Y, Zahran MH, Harraz AM, Mashaly M, Kamal AI, Ali-El-Dein B. Utility of Pre-Transplant Bladder Cycling for Patients With a Defunctionalized Bladder. A Randomized Controlled Trial. Urology. 2023 Apr;174:172-178. doi: 10.1016/j.urology.2023.01.008. Epub 2023 Jan 19. PMID 36682701
- See also: Related Info — https://www.mims.com/hongkong/news-updates/topic/bladder-cycling-pretransplant-offers-no-clinical-advantage-in-patients-with-defunctionalized-bladder

DOCUMENTS (1):
  • Study Protocol (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT06787092/Prot_000.pdf